CLINICAL TRIAL: NCT06077747
Title: Lumbar Vein Embolization for the Treatment of Chronic Headache in Patients With Nutcracker Physiology and Retrograde Lumbar Vein Flow With Epidural Venous Plexus Enhancement
Brief Title: Lumbar Vein Embolization for Chronic Headaches With Nutcracker Physiology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Zlatko Devcic, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-004668
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Chronic Headache; Nutcracker Phenomenon, Renal; Nutcracker Syndrome, Renal
MeSH Terms: conditions — Headache Disorders; Renal Nutcracker Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coil embolization of lumbar vein (Experimental): Subjects with confirmed Nutcracker physiology, retrograde lumbar vein flow, and epidural venous plexus congestion with a high pressure headache will have coil embolization of the lumbar vein.
  Interventions: Procedure: Coil Embolization of the Lumbar Vein

INTERVENTIONS:
Procedure: Coil Embolization of the Lumbar Vein — Catheter based venography will first confirm Nutcracker physiology with retrograde lumbar vein flow and epidural venous plexus congestion. The lumbar vein will then be coil embolized.

SUMMARY:
The purpose of this research is to gather information on the safety and feasibility of coiling the lumbar vein for the treatment of chronic headaches in patients with Nutcracker physiology and retrograde lumbar vein flow with epidural venous plexus congestion. All patients are extensively evaluated by a headache trained Neurologist confirming high pressure headache refractory to other treatments.

DETAILED DESCRIPTION:
This is a feasibility, non-randomized, non-blinded clinical trial enrolling patients who are at least 18 years of age for the treatment of chronic headache in the setting of Nutcracker physiology with retrograde lumbar vein flow and epidural venous plexus enhancement.

Patients are initially evaluated by a fellowship trained headache neurologist to obtain a detailed headache history, VAS score, MIDAS score, and physical examination. They are also evaluated by a neuro ophthalmologist with fundoscopic examination to assess for disc edema. A lab work-up is performed including complete blood count, basic metabolic panel, and microscopic urinalysis. A lumbar puncture and imaging work-up are then obtained as well.

Patients will proceed to an MRI to evaluate for Nutcracker physiology, retrograde lumbar vein flow, and epidural venous plexus enhancement if they meet the following criteria:

1. Daily headache from onset lasting > 3 months
2. Headache described as pressure sensation
3. Headache worsened in the Trendelenburg position
4. MRI, MRA head and neck and MR venogram negative for possible secondary causes of headache including space occupying lesions, Chiari malformation, cerebral vein thrombosis, hydrocephalus, dissection, aneurysm etc

   a. Transverse sinus stenosis is allowed to proceed
5. Exposed to CSF pressure/volume lowering medications

   a. Tried 2 of 4 unless contraindications: acetazolamide, methazolamide, indomethacin SR or spironolactone) or CSF volume removal via LP with positive or neutral response
6. Failed at least 3 typical headache preventative medications from different classes: antidepressants, antiepileptic, and blood pressure If these criteria are met, they will undergo an MRI to evaluate for Nutcracker physiology, retrograde lumbar vein flow, and epidural venous plexus enhancement. For those patients that demonstrate Nutcracker physiology with retrograde lumbar vein flow and EVP enhancement they would be eligible for the clinical trial.

If they are interested in the clinical trial, they will be evaluated in clinic by a fellowship trained interventional radiologist to review the following:

1. Procedural sedation: moderate sedation versus general anesthesia
2. Prior contrast allergies
3. Consent for procedure
4. Prior to venography the patient is taken off all headache medications for 4 weeks.

For patients that are still eligible and interested they will proceed with venography. Venography involves an evaluation of the left renal vein and left lumbar vein to confirm the findings on the MRI. If catheter-based venography confirms Nutcracker physiology with retrograde lumbar vein flow and epidural venous plexus enhancement they will then enter the clinical trial. Embolization of the lumbar vein will be performed. A follow-up venogram will then be performed to ensure there is no further retrograde lumbar vein flow.

After the embolization patient's will be followed for symptom evaluation at 1,3,7,14, and 28 days after the procedure and then monthly. They will also have a follow-up physical examination at 1 month, 3 months, 6 months and then every 6 months post-procedure. They will be followed for a total of 18 months. Some patients may need follow-up laboratory work-up and MRI post-procedure as standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Daily headache from onset lasting > 3 months.
* Headache described as pressure sensation.
* Headache worsened in the Trendelenburg position.
* Exposed to CSF pressure/volume lowering medications.
* Tried 2 of 4 unless contraindications: acetazolamide, methazolamide, indomethacin SR or spironolactone) or CSF volume removal via LP with positive or neutral response.
* Failed at least 3 typical headache preventative medications from different classes-antidepressants, antiepileptic, blood pressure medications.
* MRI demonstrates that Nutcracker physiology is present.
* Decreased SMA angle, renal vein narrowing, decreased AMD.
* Retrograde lumbar vein flow and early EVP enhancement.
* Ability to understand study procedures and to comply with them for the entire length of the study.
* Negative pregnancy test.

Exclusion Criteria:

* Evidence of disc edema.
* Positive urinalysis for hematuria or proteinuria.
* Abnormal CBC or CMP.
* MRI, MRA head and neck and MR venogram with a possible secondary causes of headache including space occupying lesions, Chiari malformation, cerebral vein thrombosis, hydrocephalus, dissection, aneurysm etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in headache pain | 1,3,7,14, and 28 days after the procedure and then monthly for 17 months
  Measured by a visual analogue scale (VAS) where 0 = no pain, 5= moderate pain, 10= worst pain
Change in Migraine Disability Assessment | 1,3,7,14, and 28 days after the procedure and then monthly for 17 months
  Measured by the Migraine Disability Assessment Test

SECONDARY OUTCOMES:
Adverse Events | 1,3,7,14, and 28 days after the procedure and then monthly for 17 months
  Number of adverse events defined as any unwanted symptom that occurred from embolizing the lumbar vein such as flank pain, proteinuria, hematuria, or pelvic congestion.
Serious Adverse Events | 1,3,7,14, and 28 days after the procedure and then monthly for 17 months
  Number of serious adverse events defined as any serious unexpected complication during or after the embolization that would result in death, is life threatening, requires prolonged hospitalization, causes persistent or significant disability or incapacity, or another condition that represents significant hazards.

CONTACTS AND LOCATIONS:
Overall Officials: Zlatko Devcic, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials